CLINICAL TRIAL: NCT05348772
Title: A First-In-Human Phase 1b, Open-Label Trial to Evaluate Safety and Tolerability of a Novel Somatic Cell Therapy, AmnioPul-02,in Subjects With Confirmed COVID-19 or Other Viral Lower Respiratory Tract Infections
Brief Title: A First-In-Human Phase 1b Study of AmnioPul-02 in COVID-19 / Other LRTI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amniotics AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AmnioPul-02-001
Record Dates: First submitted 2022-04-26; First posted 2022-04-27 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Sequential Cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AmnioPul-02 Dose level 1 (Active Comparator): AmnioPul-02 Dose level 1
  Interventions: Drug: AmnioPul-02
- AmnioPul-02 Dose level 2 (Active Comparator): AmnioPul-02 Dose level 2
  Interventions: Drug: AmnioPul-02

INTERVENTIONS:
Drug: AmnioPul-02 — Mesenchymal stem / stromal cells, MSC

SUMMARY:
This is a first-in-human (FIH), Phase 1b, open-label, dose-escalation, safety trial consisting of 3 dose levels. Subjects will always be treated in cohorts of size 3, with from 3 up to 6 cohorts i.e. 9-18 subjects.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1b, open-label, dose-escalation, safety trial consisting of 3 dose levels. Subjects will always be treated in cohorts of size 3. After a minimum safety follow-up of 7 days of the last subject in each of the cohorts where a higher dosing level may be introduced, a decision on whether to escalate, de-escalate, or stay at the current dose will be taken considering safety and efficacy data from all subjects who have been treated at the current dose level. The trial design is an adapted version of the i3+3 design and will apply 3 dose levels to separate cohorts of 3 subjects. The trial will be restricted with respect to a maximum of 9 subjects to be exposed within a dose level, and a maximum of 18 subjects to be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 to ≤80 years of age with a diagnosis of moderate or severe COVID-19, with or without pneumonia, as follows:

   1. SARS-CoV-2 infection, as confirmed by RT-PCR test within 72 hours before dosing.
   2. Subjects hospitalised primarily due to COVID-19, with symptoms considered typical for COVID-19 (eg, fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, shortness of breath, or dyspnoea requiring oxygen treatment).
   3. A score of 4, 5, or 6 on the NIAID 8-point ordinal scale for COVID-19 severity, as follows (Beigel et al 2020, Appendix II):

   i. Score 4: Hospitalised, not requiring supplemental oxygen, but requiring ongoing medical care (related to COVID-19 or to other medical conditions). ii. Score 5: Hospitalised, requiring any supplemental oxygen. iii. Score 6: Hospitalised, requiring non-invasive ventilation or use of high-flow oxygen devices.
2. Willing and able to give written informed consent prior to the initiation of any trial procedure.
3. For females only: At the time of enrolment, negative beta human chorionic gonadotropin (β-hCG) pregnancy test (serum) for women of childbearing potential (WOCBP). A woman will be considered WOCBP following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

   A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
4. If the subject is a WOCBP, must agree to practice highly effective method of contraception from screening visit and until 30 days after the last investigational medicinal product (IMP) administration. Highly effective methods of contraception include: a. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: i. Oral ii. Intravaginal iii. Transdermal b. Progestogen-only hormonal contraception associated with inhibition of ovulation: i. Oral ii. Injectable iii. Implantable c. Intrauterine devices d. Intrauterine hormone-releasing system e. Bilateral tubal occlusion f. Vasectomized partner g. Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments. The reliability of sexual abstinence needs to be evaluated in relation to the preferred and usual lifestyle of the subject) Note: Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective contraceptive methods.

Exclusion Criteria:

1. Is currently participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment in this trial (subjects who are in a follow-up period of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent).
2. Life expectancy <72 hours, in the opinion of the Investigator.
3. Subjects requiring invasive mechanical ventilation or ECMO.
4. Subjects on non-invasive CPAP ventilation or HFNO (score 6 of the NIAID 8-point ordinal scale for COVID-19 severity; Beigel et al 2020, Appendix II) are allowed, but will be excluded if they have moderate to severe ARDS (eg, same day ratio of arterial partial pressure of oxygen to fraction of inspired oxygen [PaO2/FiO2] ≤200 mmHg; or oxygen saturation [SpO2]/FiO2 ≤232 if arterial blood gas test is not available).
5. Active known cancer disease, except subjects with nonaggressive cancers such as basal cell carcinoma, or cervical carcinoma in situ.
6. Clinical evidence of active infection, in addition to the SARS-CoV-2 infection, including influenza.
7. Body weight >120 kg.
8. Pregnant or breastfeeding female subject.
9. Alzheimer's disease or dementia or any other medical condition that, in the opinion of the investigator, impact the subject's capability to properly consent with trial participation or to comply with trial protocol procedures.
10. Signs of disseminated intravascular coagulation as per the investigator's medical judgement based on the symptoms of the subject, such as unexplained bleeding, along with subject's laboratory parameters including platelet count, prothrombin time-international normalised ratio (PT-INR), partial thromboplastin time (PTT), plasma fibrinogen, and plasma D-dimer.
11. Creatinine clearance <30 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equations.
12. Abnormal liver chemistry, defined as ALT or aspartate aminotransferase (AST) or total bilirubin or PT-INR >1.5 × upper limit of normal (ULN).
13. Severe cardiovascular diseases (severe or unstable angina, congestive heart failure (New York Heart Association [NYHA] III-IV), myocardial infarction within past 1 year, uncontrolled hypertension, and uncontrolled arrhythmia).
14. Electrocardiogram (ECG) findings with corrected QT interval using Fridericia's (QTcF) formula >500 msec.
15. Subjects with a known or suspected hypersensitivity to MSCs or contaminants (DMSO and Accutase).
16. COVID-19 vaccine administered within less than 14 days prior to screening.
17. Known thrombosis or thromboembolic event (TEE) or known medical history of TEEs (eg, cerebrovascular accidents, transient ischemic attack, myocardial infarction, pulmonary embolism, and deep vein thrombosis) within the previous 3 months or those subjects particularly at risk for TEEs (eg, history of thrombophilia, permanent immobilisation, or permanent paralysis of their lower extremities).
18. Any other medical condition which, in the opinion of the investigator, would impact the safety of the subject or interfere with the subject's ability to comply with the trial and follow-up procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting adverse events/toxicities (DLTs) | Day 7
  The primary endpoint is the number of subject dose-limiting adverse events/toxicities (DLTs) associated with administration of AmnioPul-02 at each dose level.

SECONDARY OUTCOMES:
OS | Day 22
  Overall survival defined as time from ATIMP infusion to death for any cause
Event-free survival | Day 22
  Event-free survival (defined as time from ATIMP infusion to "event" or death)
Ventilator-free days | Day 22
  Ventilator-free days defined as days alive and free from mechanical ventilation
Time to clinical response | Day 22
  Time to clinical response defined as time from ATIMP infusion to improvement of at least 1 point in the National Institute of Allergy and Infectious Diseases (NIAID) 8-point ordinal scale for COVID-19 severity
OS | 1 year
  Overall survival defined as time from ATIMP infusion to death for any cause
Time to hospital discharge | Day 22
  Time to hospital discharge defined as time from ATIMP infusion to time to hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Infection clinic, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No